CLINICAL TRIAL: NCT05097820
Title: Prospective Observational Study on SEBBIN Silicone Gel-filled Testicular Implants
Status: Recruiting | Type: Observational
Sponsor: University Hospital, Ghent (Other)
Collaborators: Groupe SEBBIN (Industry)
Responsible Party: Sponsor
Other Study IDs: BC-8299
Record Dates: First submitted 2021-09-21; First posted 2021-10-28 (Actual); Last update posted 2024-09-19 (Actual); Status verified 2024-09

CONDITIONS: Testicular Cancer; Testicular Torsion; Gender Dysphoria; Undescended Testes; Orchitis; Testicular Agenesis; Testicular Atrophy; Prosthesis Durability
Keywords: testicular prosthesis
MeSH Terms: conditions — Testicular Neoplasms; Spermatic Cord Torsion; Gender Dysphoria; Cryptorchidism; Orchitis; Anorchia; Prosthesis Failure

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 2 Years
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- Cisgender patients: All cisgender patients in which one or two testicular prostheses are to be implanted for various reasons.
  Interventions: Device: Placement of testicular prosthesis
- Transgender patients: All transgender patients in which one or two testicular prostheses are to be implanted for gender reassignment surgery.
  Interventions: Device: Placement of testicular prosthesis

INTERVENTIONS:
Device: Placement of testicular prosthesis — The surgical implantation of one or two testicular prostheses on request of the patient

SUMMARY:
To analyze the short and long term postoperative clinical outcome and patient satisfaction of silicone gel-filled testicular implants.

DETAILED DESCRIPTION:
Testicular implants made from various materials have been in use since 1941. The lack of a testicle has proven to be a psychologically traumatic experience for men of all ages. Therefore, testicular implants are placed in the scrotum for various reasons on request of the patient.The intended target population for the silicone gel-filled testicular implants of Groupe SEBBIN is any patient (children or adults) with agenesis or testicular atrophy, undescended testicle, testicular tumour, epididymitis / orchitis, or a trauma, for whom an orchidectomy with placement of a testicular prosthesis is indicated. Testicular implants are also indicated for sex reassignment surgeries.

The main complications after testicular implant placement recorded in the literature include extrusion, scrotal contraction, pain, hematoma, and infection. The literature about testicular implant is sparse, and no report on the use of SEBBIN silicone gel-filled testicular implants have been identified in the scientific literature.

The Gel-filled Testicular Implant medical devices are manufactured by GROUPE SEBBIN under the brand name 'Laboratoires SEBBIN'. The Gel-filled Testicular Implant medical devices are presented sterile (Ethylene oxide sterilization) and are double wrapped for single use.

The medical grade raw materials used for the manufacturing of these prostheses are bio-compatible and completely traceable. The substances belong to the polydimethylsiloxane family.

This study is part of the clinical evaluation of SEBBIN silicone gel-filled testicular implants, included in the technical file of the device. The aim of the study is to gather data on the safety and effectiveness of the device. For this purpose, the overall short and long term complication rate and complication grade. Secondly, the investigators evaluate patient satisfaction and quality of life by use of questionnaires

ELIGIBILITY:
Inclusion Criteria:

* The patient is an adult or a child at the time of testicular implant placement.
* The patient is a candidate to unilateral or bilateral testicular implant placement.
* The patient has been informed of the study, has read the patient information letter and provided oral and written consent.
* If the patient is of French nationality, he/she must be affiliated to the French Social Security.

Exclusion Criteria:

* The patient has silicone implants somewhere else than in the scrotal sac (except for a penile prosthesis).
* The patient was diagnosed with one of the following pathologies:

Systemic lupus erythematous, Sjogren syndrome, scleroderma, polymyositis, or any other connective tissue disease.

Rheumatoid arthritis, crystalline arthritis, infectious arthritis, spondyloarthropathies, or any other inflammatory arthritic disease.

Arthritis, fibromyalgia, chronic fatigue syndrome, or any other mechanic or degenerative non-inflammatory rheumatic disease.

The patient has any other underlying condition that could delay healing.

- Custom-designed implants are used for surgery.

Ages: 0 Years to 110 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Any undividual with an underlying reason for testicular loss with a specific wish for testicular implant placement.
  Any patient with the underlying condidion of gender dysphoria with the specific wish for testicular implant placement as a form of gender reassignment surgery.
Sampling Method: Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2021-02-05 (Actual); Primary Completion 2030-12-31 (Estimated); Study Completion 2030-12-31 (Estimated)

PRIMARY OUTCOMES:
Short term complication rate | Within 90 days postoperatively
  Cathegorized according to Clavien-Dindo Classification
Long term complication rate | At 2 years of follow-up
  Desciption of overall complications related to testicular prosthesis placement.

SECONDARY OUTCOMES:
Change in self-esteem scoring | Baseline questionnaire, followed by reassessment at 3, 6, 12 and 24 months of follow-up
  Assessed by the Rosenberg Self-Esteem Scale (strongly disagree - strongly agree)
Body image of scrotum | Baseline questionnaire, followed by reassessment at 3, 6, 12 and 24 months of follow-up
  Assessed with non-validated likert scale quationnaires
Satisfaction with prosthesis | Baseline questionnaire, followed by reassessment at 3, 6, 12 and 24 months of follow-up
  Assessed with non-validated likert scale quationnaires

CONTACTS AND LOCATIONS:
Overall Officials: Anne-Françoise Spinoit, MD, PhD, Principal Investigator — University Hospital, Ghent
Locations (1):
- University Hospital Ghent, Ghent, East-Flanders, Belgium

IPD SHARING:
Plan to Share IPD: Undecided
After publication of findings, the individual patient data can be provided upon request.